CLINICAL TRIAL: NCT06246682
Title: The Impact of Mastoid Condition and Ossicular Reconstruction on the Outcome of the Transcanal Endoscopic Management of Localized Atticoantral Cholesteatoma Patients
Brief Title: Impact of Mastoid Condition on Results of Endoscopic Management of Cholesteatoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Farghaly Abdelrahman Mekki, Assistant lecturer of otolaryngology sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-01-03MD
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Cholesteatoma of Attic; Cholesteatoma, Middle Ear
Keywords: cholesteatoma; Endoscopic ear surgery; mastoid process
MeSH Terms: conditions — Cholesteatoma, Middle Ear; Cholesteatoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cholesteatoma removal by otoendoscope (Other): removal of the cholesteatoma in atticoantral region by otoendoscope
  Interventions: Procedure: Transcanal Endoscopic removal of atticoantral cholesteatoma

INTERVENTIONS:
Procedure: Transcanal Endoscopic removal of atticoantral cholesteatoma — removal of the cholesteatoma presented in the atticoantral region by otoendoscope

SUMMARY:
The goal of this interventional study is to learn about the effect of mastoid process status and the method of ossicular reconstruction on the results of the procedure transcanal endoscopic management of patients with localized atticoantral cholesteatoma

DETAILED DESCRIPTION:
Acquired cholesteatoma is a special form of chronic otitis media in which keratinizing squamous epithelium grows from the tympanic membrane or/and the auditory canal skin into the middle ear mucosa. Acquired cholesteatomas of the middle ear are further divided into primary acquired and secondary acquired forms. The primary acquired cholesteatoma is the most frequent type of acquired cholesteatoma and develops by the progression of an initial retraction pocket into a cholesteatoma. Primary acquired cholesteatomas are named relative to the site of the pocket origin: (1) attic cholesteatoma consecutive to a pars flaccida pocket,(2) mesotympanic cholesteatoma due to a pars tensa pocket, and (3) combined forms, due to double pockets. The predominant form of acquired cholesteatoma in children develops in 80% from retraction pockets of the pars tensa whereas in adults, this form develops mainly in the pars flaccida.

The diagnosis of cholesteatoma is made on otoscopic examination, including endoscopic and microscopic evaluation, imaging, or surgical exploration. The symptoms of cholesteatoma vary; some cholesteatomas are asymptomatic, whereas others become infected and rapidly cause bone destruction. Some patients will present with slowly progressive conductive hearing loss and, frequently, with chronic otitis and purulent otorrhea. The otorrhea from an infected cholesteatoma often is malodorous because of the frequent infection with anaerobic bacteria. Some patients will have signs and symptoms of the complications of a cholesteatoma: vertigo and hearing loss caused by a labyrinthine fistula, facial nerve paralysis, or intracranial infection.

there are some contraindications to the use of exclusively endoscopic approaches. For example, if cholesteatoma involves the mastoid cavity, it is not possible to control and remove it by only a transcanal approach; the use of the microscope in combination with the endoscope is recommended. Also, a narrow external ear canal, or external ear malformation, can pose general anatomical difficulties for exclusively endoscopic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with primary acquired localized atticoantral cholesteatoma.

Exclusion Criteria:

* Age group: patients below 12 years old.
* Patients presenting with congenital or secondary acquired cholesteatoma.
* Patients presenting with extensive, residual, or recurrent cholesteatoma.
* Patients with craniofacial anomalies.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
recurrence of cholesteatoma after procedure according to mastoid condition | six months postoperative after the procedure
  measurement of changes in recurrence rate of cholesteatoma after its removal according to different types of mastoid process

CONTACTS AND LOCATIONS:
Overall Officials: farghali Abdelrahman, Principal Investigator — Sohag University
Locations (1):
- faculty of medicine Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchioni D, Piccinini A, Alicandri-Ciufelli M, Presutti L. Endoscopic anatomy and ventilation of the epitympanum. Otolaryngol Clin North Am. 2013 Apr;46(2):165-78. doi: 10.1016/j.otc.2012.10.002. Epub 2012 Nov 27. PMID 23566903
- [Background] Presutti L, Anschuetz L, Rubini A, Ruberto M, Alicandri-Ciufelli M, Dematte M, Caversaccio M, Marchioni D. The Impact of the Transcanal Endoscopic Approach and Mastoid Preservation on Recurrence of Primary Acquired Attic Cholesteatoma. Otol Neurotol. 2018 Apr;39(4):445-450. doi: 10.1097/MAO.0000000000001712. PMID 29342049